CLINICAL TRIAL: NCT01027364
Title: B-LONG: An Open-Label, Multicenter Evaluation of the Safety, Pharmacokinetics, and Efficacy of Recombinant, Long-acting Coagulation Factor IX Fc Fusion Protein (rFIXFc) in the Prevention and Treatment of Bleeding in Previously Treated Subjects With Severe Hemophilia B
Brief Title: Study of Recombinant Factor IX Fc Fusion Protein (rFIXFc) in Participants With Hemophilia B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ Therapeutics Inc. (Industry)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 998HB102; 2009-014295-21 (EudraCT Number)
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2018-08

CONDITIONS: Severe Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fixed Weekly Interval (Experimental): 50 IU/kg rFIXFc via intravenous (IV) injection once every 7 days initially, then at a dose indicated by the participant's baseline pharmacokinetic (PK) assessment that ensured a target trough of 1% to 3% above baseline or higher, as clinically indicated. Adjustments to the initial weekly dose of rFIXFc (50 IU/kg) were to be made based on baseline PK assessments, occurrence of spontaneous bleeding episodes, and the trough levels, which were to be monitored at Weeks 4, 16, 26, and 39.
  Prior to the first dose of rFIXFc, participants in the Sequential PK subgroup were to receive a single dose of 50 IU/kg BeneFIX administered IV in the clinic, followed by PK sampling. A single dose of 50 IU/kg rFIXFc was administered following a 120-hour washout from BeneFIX, followed by PK sampling for a baseline PK profiling. At Week 26 (±1 week) subjects were to receive a single dose of 50 IU/kg rFIXFc for repeat PK profiling.
  Interventions: Drug: Factor IX (rFIXFc); Drug: rFIX
- Individualized Interval (Experimental): 100 IU/kg rFIXFc via IV injection once every 10 days initially, then at an interval derived from the baseline PK assessment that ensured a target trough of 1% to 3% above baseline or higher, as clinically indicated. Adjustments to the initial 10-day interval were to be made based on baseline PK assessments and trough levels, which were monitored at Weeks 4, 16, 26, and 39.
  Interventions: Drug: Factor IX (rFIXFc)
- On Demand (Experimental): 20 to 100 IU/kg rFIXFc via IV injection, or the dose indicated by the participant's baseline PK to target a plasma level of 20% to 100%, as needed for the treatment of mild to severe bleeding episodes
  Interventions: Drug: Factor IX (rFIXFc)
- Surgery (Experimental): The surgical period and dosing are dependent on the type of surgery the participant undergoes. Participants who started the study in one of the other treatment arms prior to surgery will return to the original treatment arm. Participants who joined the study in the Surgery arm will be assigned to one of the other treatment arms following post-operative rehabilitation.
  Interventions: Drug: Factor IX (rFIXFc)

INTERVENTIONS:
Drug: Factor IX (rFIXFc)
  Other Names: Recombinant Human Factor IX Fc Fusion Protein
Drug: rFIX
  Other Names: Recombinant Factor IX; BeneFIX®
  Arms: Fixed Weekly Interval

SUMMARY:
The primary objectives of the study were: to evaluate the safety and tolerability of rFIXFc; to evaluate the efficacy of rFIXFc in all treatment arms; to evaluate the effectiveness of prophylaxis over on-demand (episodic) therapy by comparing the annualized number of bleeding episodes between participants receiving rFIXFc on each prevention (prophylaxis) regimen and participants receiving rFIXFc on an episodic regimen. The secondary objectives of the study were: to evaluate and assess the pharmacokinetic (PK) parameter estimates of rFIXFc and rFIX (BeneFIX®) at baseline in the Sequential PK subgroup as well as rFIXFc at Week 26 (±1 week); to evaluate participants' response to treatment; to evaluate rFIXFc consumption.

ELIGIBILITY:
Inclusion Criteria:

* Male and 12 years of age and older and weigh at least 40 kg
* Diagnosed with hemophilia B (baseline Factor IX level less than or equal to 2%)
* History of at least 100 exposure days to any Factor IX product
* Platelet count ≥100,000 cells/μL

Exclusion Criteria:

* History of Factor IX inhibitors
* Kidney or liver dysfunction
* Diagnosed with another coagulation defect other than hemophilia B
* Prior history of anaphylaxis associated with any Factor IX or intravenous (IV) immunoglobulin administration

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2009-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Bioverativ Therapeutics Inc.
Locations (51):
- United States (9):
  - Research Site, Phoenix, Arizona
  - Research Site, Sacramento, California
  - Research Site, Aurora, Colorado
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, East Lansing, Michigan
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Seattle, Washington
- Australia (3):
  - Research Site, Camperdown, New South Wales
  - Research Site, Adelaide, South Australia
  - Research Site, Perth, Western Australia
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Leuven
- Research Site, Campinas, Brazil
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Vancouver
- China (4):
  - Research site, Beijing
  - Research Site, Guangzhou
  - Research Site, Shanghai
  - Research Site, Tianjin
- France (2):
  - Research Site, Lyon
  - Research Site, Marseille
- Germany (2):
  - Research Site, Berlin
  - Research Site, Bonn
- Hong Kong (2):
  - Research Site, Pokfulam
  - Research Site, Shatin
- India (4):
  - Research Site, Ludhiana, Punjab
  - Research Site, Vellore, Tamil Nadu
  - Research Site, Bangalore
  - Research Site, Pune
- Italy (2):
  - Research Site, Florence
  - Research Site, Milan
- Japan (6):
  - Research Site, Kasihara-City
  - Research Site, Kawasaki
  - Research Site, Kitakyushu
  - Research Site, Nagoya
  - Ressearch Site, Suginami-ku
  - Research Site, Tokyo
- Poland (2):
  - Research Site, Lodz
  - Research Site, Warsaw
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Africa (2):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Cape Town, Western Cape
- Sweden (2):
  - Research Site, Malmo
  - Research Site, Stockholm
- United Kingdom (2):
  - Research Site, Cambridge
  - Research Site, London

REFERENCES:
- [Result] Powell JS, Pasi KJ, Ragni MV, Ozelo MC, Valentino LA, Mahlangu JN, Josephson NC, Perry D, Manco-Johnson MJ, Apte S, Baker RI, Chan GC, Novitzky N, Wong RS, Krassova S, Allen G, Jiang H, Innes A, Li S, Cristiano LM, Goyal J, Sommer JM, Dumont JA, Nugent K, Vigliani G, Brennan A, Luk A, Pierce GF; B-LONG Investigators. Phase 3 study of recombinant factor IX Fc fusion protein in hemophilia B. N Engl J Med. 2013 Dec 12;369(24):2313-23. doi: 10.1056/NEJMoa1305074. Epub 2013 Dec 4. PMID 24304002
- [Derived] Shapiro AD, Kulkarni R, Ragni MV, Chambost H, Mahlangu J, Oldenburg J, Nolan B, Ozelo MC, Foster MC, Willemze A, Barnowski C, Jain N, Winding B, Dumont J, Lethagen S, Barnes C, Pasi KJ. Post hoc longitudinal assessment of the efficacy and safety of recombinant factor IX Fc fusion protein in hemophilia B. Blood Adv. 2023 Jul 11;7(13):3049-3057. doi: 10.1182/bloodadvances.2022009230. PMID 36848635

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Weekly Prophylaxis: 50 IU/kg rFIXFc via intravenous (IV) injection once every 7 days initially, then at a dose indicated by the participant's baseline pharmacokinetic (PK) assessment that ensured a target trough of 1% to 3% above baseline or higher, as clinically indicated. Adjustments to the initial weekly dose of rFIXFc (50 IU/kg) were to be made based on baseline PK assessments, occurrence of spontaneous bleeding episodes, and the trough levels, which were to be monitored at Weeks 4, 16, 26, and 39.
  Prior to the first dose of rFIXFc, participants in the Sequential PK subgroup were to receive a single dose of 50 IU/kg BeneFIX administered IV in the clinic, followed by PK sampling. A single dose of 50 IU/kg rFIXFc was administered following a 120-hour washout from BeneFIX, followed by PK sampling for a baseline PK profiling. At Week 26 (±1 week) subjects were to receive a single dose of 50 IU/kg rFIXFc for repeat PK profiling.
- Arm 2: Individualized Interval Prophylaxis: 100 IU/kg rFIXFc via IV injection once every 10 days initially, then at an interval derived from the baseline PK assessment that ensured a target trough of 1% to 3% above baseline or higher, as clinically indicated. Adjustments to the initial 10-day interval were to be made based on baseline PK assessments and trough levels, which were monitored at Weeks 4, 16, 26, and 39.
- Arm 3: Episodic (On Demand): 20 to 100 IU/kg rFIXFc via IV injection, or the dose indicated by the participant's baseline PK to target a plasma level of 20% to 100%, as needed for the treatment of mild to severe bleeding episodes
- Arm 4: Perioperative Management: The surgical period and dosing were dependent on the type of surgery the participant underwent. Participants who started the study in one of the other treatment arms prior to surgery returned to the original treatment arm. Participants who joined the study in the Surgery arm were assigned to one of the other treatment arms following post-operative rehabilitation.
Period: Overall Study
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand) | Arm 4: Perioperative Management
Started | 63 | 29 | 27 | 4 (12 total participants in Arm 4 (6 started in Arm 4; 5 joined from Arm 1; 1 joined from Arm 3))
Enrolled in Sequential PK Subgroup | 22 | 0 | 0 | 0
Joined Arm 4 for Surgery Then Returned | 5 | 0 | 1 | 0
Started Arm 4 Then Joined Another Arm | 2 | 0 | 0 | 0
Completed | 59 | 27 | 26 | 3 (11 participants total completed Arm 4 (3: compl. Arm 4 only; 7: cont. to Arm 1; 1: cont. to Arm 3))
Not Completed | 4 | 2 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand) | Arm 4: Perioperative Management | Total
Number analyzed (Participants) | 63 | 29 | 27 | 4 | 123
Age, Continuous [Median (Full Range); unit: years] — The 4 participants represented in the Perioperative Management arm includes participants who were enrolled in this arm only. A total of 12 participants underwent 14 major surgeries in this study, and 8 participants either joined this arm from another arm, or who started this arm, then joined another arm (see Participant Flow milestones for details).
  years | 28.0 [12 to 71] | 33.0 [12 to 62] | 36.0 [14 to 64] | 40.5 [30 to 61] | 30.0 [12 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 63 | 29 | 27 | 4 | 123

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities
Description: Clinical laboratory evaluations included hematology and blood chemistry. Table does not include laboratory tests evaluated during the surgical/rehabilitation period. Because the perioperative management period represents a unique clinical situation, safety data obtained during the surgical/rehabilitation period for participants in Arm 4 were included in listings and reviewed separately. Review of the listing was sufficient to assess this endpoint. ULN=upper limit of normal.
Time Frame: up to 52 weeks ± 1 week
Population: Safety Analysis Set: participants who received at least 1 dose of BeneFIX or rFIXFc; n=the number of participants with at least one post-baseline value. For this study, a table was not generated for potentially clinically significant laboratory abnormalities for participants in the perioperative management/surgical arm (Arm 4).
Measure: Number; unit: participants
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 63 | 29 | 27
participants
  White Blood Cells <3.0*10^9/L; n=62, 28, 27 | 2 | 0 | 2
  White Blood Cells >=16*10^9/L; n=62, 28, 27 | 0 | 0 | 0
  Lymphocytes <0.8*10^9/L; n=60, 28, 26 | 1 | 2 | 3
  Lymphocytes >12*10^9/L; n=60, 28, 26 | 0 | 0 | 0
  Neutrophils <1.5*10^9/L; n=60, 28, 26 | 2 | 0 | 1
  Neutrophils >13.5*10^9/L; n=60, 28, 26 | 0 | 0 | 0
  Monocytes >2.5*10^9/L; n=60, 28, 26 | 0 | 0 | 0
  Eosinophils >1.6*10^9/L; n=60, 28, 26 | 0 | 0 | 0
  Basophils >1.6*10^9/L; n=60, 28, 26 | 0 | 0 | 0
  Red Blood Cells <=3.5*10^12/L; n=62, 28, 27 | 1 | 0 | 0
  Red Blood Cells >=6.4*10^12/L; n=62, 28, 27 | 0 | 0 | 0
  Hemoglobin <=115 g/L; n=62, 28, 27 | 1 | 0 | 0
  Hemoglobin >=190 g/L; n=62, 28, 27 | 0 | 0 | 0
  Hematocrit <=37%; n=62, 28, 27 | 4 | 0 | 2
  Hematocrit >=60%; n=62, 28, 27 | 0 | 0 | 0
  Platelets <=75*10^9/L; n=62, 28, 27 | 0 | 0 | 1
  Platelets >=700*10^9/L; n=62, 28, 27 | 0 | 0 | 0
  Alanine Aminotransferase >=3*ULN; n=62, 28, 27 | 0 | 0 | 2
  Aspartate Aminotransferase >=3*ULN; n=62, 28, 27 | 2 | 1 | 1
  Alkaline Phosphatase >=3*ULN; n=62, 28, 27 | 0 | 0 | 0
  Total Bilirubin >=34.2 µmol/L; n=62, 28, 27 | 1 | 0 | 0
  Blood Urea Nitrogen >=10.7 mmol/L; n=62, 28, 27 | 1 | 0 | 0
  Creatinine >=176.8 µmol/L; n=62, 28, 27 | 1 | 0 | 0
  Sodium <=126 mmol/L; n=62, 28, 27 | 0 | 0 | 0
  Sodium >=156 mmol/L; n=62, 28, 27 | 0 | 0 | 0
  Potassium <=3 mmol/L; n=62, 28, 27 | 0 | 0 | 0
  Potassium >=6 mmol/L; n=62, 28, 27 | 0 | 0 | 0
  Chloride <=90 mmol/L; n=62, 28, 27 | 0 | 0 | 0
  Chloride >=118 mmol/L; n=62, 28, 27 | 0 | 0 | 0
  Phosphate <=0.55 mmol/L n=62, 28, 27 | 0 | 0 | 1
  Phosphate >=1.71 mmol/L; n=62, 28, 27 | 1 | 1 | 0
  Glucose <=2.22 mmol/L; n=62, 28, 27 | 0 | 0 | 0
  Glucose >=9.71 mmol/L; n=62, 28, 27 | 4 | 1 | 0
  Albumin <=25 g/L; n=62, 28, 27 | 0 | 0 | 0
  Total Protein <=45 g/L; n=62, 28, 27 | 0 | 0 | 0
  Total Protein >=100 g/L; n=62, 28, 27 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: AE=any untoward medical occurrence that did not necessarily have a causal relationship with this treatment, and could be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study product, whether related or not. TE=event present prior to receiving the first injection of BeneFIX or rFIXFc that subsequently worsened in severity or not present prior to receiving the first injection but subsequently appeared before last visit on study. Serious AE (SAE)=AE resulting in death, immediate risk of death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, or a congenital/anomaly/birth defect, or any other medically important event. Related=related, possibly related, and relationship missing. Data include AEs emergent during the surgical/rehabilitation period; AE data are included in each treatment arm only for the time each participant was enrolled in that arm.
Time Frame: up to 52 weeks + 30 days ± 1 week
Population: Safety Analysis Set: participants who received at least 1 dose of BeneFIX or rFIXFc. A participant may have been in more than one group (i.e., participants in Arm 4 who were also in Arm 1, 2, or 3; please see Participant Flow for details). Participants with at least one TESAE reported are included in the TEAE count.
Measure: Number; unit: participants
Groups:
- Arm 1: Weekly Prophylaxis-BeneFIX; Arm 1: Weekly Prophylaxis-rFIXFc: 50 IU/kg rFIXFc via intravenous (IV) injection once every 7 days initially, then at a dose indicated by the participant's baseline pharmacokinetic (PK) assessment that ensured a target trough of 1% to 3% above baseline or higher, as clinically indicated. Adjustments to the initial weekly dose of rFIXFc (50 IU/kg) were to be made based on baseline PK assessments, occurrence of spontaneous bleeding episodes, and the trough levels, which were to be monitored at Weeks 4, 16, 26, and 39.
  Prior to the first dose of rFIXFc, participants in the Sequential PK subgroup were to receive a single dose of 50 IU/kg BeneFIX administered IV in the clinic, followed by PK sampling. A single dose of 50 IU/kg rFIXFc was administered following a 120-hour washout from BeneFIX, followed by PK sampling for a baseline PK profiling. At Week 26 (±1 week) subjects were to receive a single dose of 50 IU/kg rFIXFc for repeat PK profiling.
Arm/Group | Arm 1: Weekly Prophylaxis-BeneFIX | Arm 1: Weekly Prophylaxis-rFIXFc | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand) | Arm 4: Perioperative Management
Number analyzed (Participants) | 23 | 63 | 29 | 27 | 12
participants
  >=1 TEAE | 2 | 45 | 23 | 20 | 10
  >=1 Related TEAE | 0 | 5 | 4 | 1 | 0
  >=1 TESAE | 0 | 5 | 4 | 4 | 3
  >=1 Related TESAE | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Non-serious Treatment-emergent Adverse Events (TEAEs) During the Surgical / Rehabilitation Period
Description: AE=any untoward medical occurrence that did not necessarily have a causal relationship with this treatment, and could be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study product, whether related or not. TEAE=AE present prior to receiving the first injection of BeneFIX or rFIXFc that subsequently worsened in severity or was not present prior to receiving the first injection but subsequently appeared before last visit on study. Participants are counted once if they report multiple events in the same system organ class (SOC) or preferred term (PT). Coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 15.0 dictionary. The following SOCs are abbreviated in the table: Immune System (IS); Injury, Poisoning, and Procedural (IPP); Metabolism and Nutrition (MN); Musculoskeletal and Connective Tissue (MCT); Respiratory, Thoracic and Mediastinal (RTM); Skin and Subcutaneous Tissue (SST).
Time Frame: up to 52 weeks + 30 days ± 1 week
Population: Safety Analysis Set: participants who received at least 1 dose of BeneFIX or rFIXFc. A participant may have been in more than one group (i.e., participants in Arm 4 who were also in Arm 1, 2, or 3; please see Participant Flow for details).
Measure: Number; unit: participants
Units Other Than Participants: Participants With At Least 1 TEAE
Arm/Group | Arm 4: Perioperative Management
Number analyzed (Participants) | 12
Number analyzed (Participants With At Least 1 TEAE) | 8
participants
  SOC: Blood/Lymphatic System Disorders; PT: Anaemia | 2
  SOC: Ear and Labyrinth Disorders; PT: Vertigo | 1
  SOC: Gastrointestinal Disorders; PT: Constipation | 1
  SOC: Gastrointestinal Disorders; PT: Nausea | 1
  SOC: Gastrointestinal Disorders; PT: Vomiting | 1
  SOC: General Disorders; PT: Asthenia | 1
  SOC: General Disorders; PT: Infusion Site Pain | 1
  SOC: IS Disorders; PT: Drug Hypersensitivity | 1
  SOC: Infections/Infestations; PT: Cellulitis | 1
  SOC: IPP Complications; PT: Incision Site Pain | 1
  SOC: IPP Complications; PT: Procedural Pain | 1
  SOC: IPP Complications; PT: Wound Complication | 1
  SOC: Investigations; PT: Weight Increased | 1
  SOC: MN Disorders; PT: Decreased Appetite | 1
  SOC: MCT Disorders; PT: Muscle Spasms | 1
  SOC: Nervous System Disorders; PT: Dizziness | 2
  SOC: Nervous System Disorders; PT: Headache | 1
  SOC: Nervous System (NS) Disorders; PT: Neuralgia | 1
  SOC: NS Disorders; PT: Neuropathy Peripheral | 1
  SOC: Psychiatric Disorders; PT: Anxiety | 1
  SOC: Psychiatric Disorders; PT: Insomnia | 1
  SOC: RTM Disorders; PT: Dyspnoea | 1
  SOC: RTM Disorders; Oropharyngeal Pain | 1
  SOC: SST Disorders; PT: Hyperhidrosis | 1
  SOC: Vascular Disorders; PT: Hypertension | 1
  SOC: Vascular Disorders; PT: Hypotension | 1

4. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs) During the Surgical / Rehabilitation Period
Description: SAE=AE resulting in death, immediate risk of death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, or a congenital/anomaly/birth defect, or any other medically important event. TESAE=SAE present prior to receiving the first injection of BeneFIX or rFIXFc that subsequently worsened in severity or was not present prior to receiving the first injection but subsequently appeared before last visit on study. Participants are counted once if they report multiple events in the same system organ class (SOC) or preferred term (PT). Coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 15.0 dictionary. The following SOC is abbreviated in the table: Injury, Poisoning, and Procedural (IPP).
Time Frame: up to 52 weeks + 30 days ± 1 week
Population: as for outcome 3
Measure: Number; unit: participants
Units Other Than Participants: Participants With At Least 1 TESAE
Arm/Group | Arm 4: Perioperative Management
Number analyzed (Participants) | 12
Number analyzed (Participants With At Least 1 TESAE) | 3
participants
  SOC: Cardiac Disorders; PT: Tachycardia | 1
  SOC: Infections/Infestations; PT: Bacterial Sepsis | 1
  SOC: Infections/Infestations; PT: Pilondial Cyst | 1
  SOC: Infections/Infestations; PT: Tooth Abscess | 1
  SOC: IPP Complications; PT: Limb Crushing Injury | 1

5. Secondary Outcome: Participant Assessment of Response to Injections to Treat a Bleeding Episode
Description: Participant's assessment of the response to the first rFIXFc injection for each bleeding episode. Percentages were based on the number of bleeding episodes for which a response was provided for the first injection, using the following 4-point scale: excellent=abrupt pain relief and/or improvement in signs of bleeding within approximately 8 hours after the initial injection; good=definite pain relief and/or improvement in signs of bleeding within approximately 8 hours after an injection, but possibly requiring more than one injection after 24 to 48 hours for complete resolution; moderate=probable or slight beneficial effect within 8 hours after the initial injection and requiring more than one injection; no response=no improvement, or condition worsened, within approximately 8 hours after the initial injection.
Time Frame: up to 52 weeks ± 1 week
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc and had a bleeding episode; participants with a non-evaluable bleeding episode are counted in the 'number of participants analyzed,' but not the percentages.
Measure: Number; unit: percentage of responses
Units Other Than Participants: Bleeding Episodes
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 47 | 15 | 27
Number analyzed (Bleeding Episodes) | 156 | 63 | 394
percentage of responses
  Excellent or Good | 78.8 | 74.6 | 87.1
  Excellent | 35.3 | 31.7 | 37.3
  Good | 43.6 | 42.9 | 49.7
  Moderate | 18.6 | 22.2 | 11.9
  No Response | 2.6 | 3.2 | 1.0

6. Secondary Outcome: Physicians' Global Assessments of Participants' Response to Treatment With rFIXFc
Description: Physicians assessed each participant's response to rFIXFc using a 4-point scale: excellent=bleeding episodes responded to less than or equal to the usual number of injections or less than or equal to the usual dose of rFIXFc, or the rate of breakthrough bleeding during prophylaxis was less than or equal to that usually observed; effective=most bleeding episodes responded to the same number of injections and dose, but some required more injections or higher doses, or there was a minor increase in the rate of breakthrough bleeding; partially effective=bleeding episodes most often required more injections and/or higher doses than expected, or adequate breakthrough bleeding prevention during prophylaxis required more frequent injections and/or higher doses; ineffective=routine failure to control hemostasis or hemostatic control required additional agents. Percentage of the total count of scale responses for all participants is presented. Multiple responses per participant are counted.
Time Frame: up to 52 weeks ± 1 week
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc, had evaluable efficacy assessments, and had nonmissing observations at time point.
Measure: Number; unit: percentage of responses
Units Other Than Participants: Responses
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 61 | 26 | 27
Number analyzed (Responses) | 267 | 123 | 96
percentage of responses
  Excellent | 74.5 | 73.2 | 58.3
  Effective | 24.3 | 26.0 | 39.6
  Partially Effective | 1.1 | 0.8 | 2.1
  Ineffective | 0 | 0 | 0

7. Secondary Outcome: Annualized rFIXFc Consumption Per Participant
Description: Consumption is calculated for the efficacy period (EP). In Arms 1 and 2, the EP started with date and time of first prophylactic dose following a completed PK sampling period and ended with last dose administered (for prophylaxis or a bleeding episode). In Arm 3, the EP started following last PK sampling timepoint and ended with either date of last contact or date of last entry into the eDiary, whichever was later. The EP was interrupted for the repeat PK period in Arm 1 (sequential PK subgroup) and for all surgical/rehabilitation periods (for both major and minor surgeries) in all 3 arms. Overall units (IU/kg) of annualized rFIXFc consumption = [Total rFIXFc IU/kg received during the EP / number of days in EP]*365.25.
Time Frame: up to 52 weeks ± 1 week (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc with evaluable data in the efficacy period. 'Overall' n=all participants in the Full Analysis Set with evaluable data in the efficacy period; 'Last 3 Months on Study' n=all participants in the Full Analysis Set with evaluable data and >=6 months on study.
Measure: Mean (Standard Deviation); unit: IU/kg rFIXFc per participant per year
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 61 | 26 | 27
IU/kg rFIXFc per participant per year
  Overall (n=61, 26, 27) | 2686.94 (825.969) | 3371.92 (649.690) | 936.70 (481.764)
  Last 3 months on study (n=58, 26, 27) | 2467.32 (978.529) | 3497.78 (957.377) | 957.73 (699.640)

8. Secondary Outcome: Average Weekly Dose For the Fixed Weekly Interval Prophylaxis Arm
Description: Average weekly dose = (total IU/kg of all eligible prophylactic doses in the included intervals / total number of days in the included intervals)*7. Eligible dose = the first of the 2 doses defining the interval. Participants could have multiple prophylactic dose changes. Prophylactic dosing = from first prophylactic injection received for rFIXFc to the last prophylactic injection on study. Intervals between 2 prophylactic doses separated by a bleed/surgery/PK visit were not included. In Arm 1, the efficacy period (EP) started with date and time of first prophylactic dose following a completed PK sampling period and ended with last dose administered (for prophylaxis or a bleeding episode). The EP was interrupted for the repeat PK period in Arm 1 (sequential PK subgroup) and for all surgical/rehabilitation periods (for both major and minor surgeries).
Time Frame: up to 52 weeks ± 1 week (efficacy period as defined in description)
Population: Full Analysis Set: participants in Arm 1 who received at least 1 dose of rFIXFc with evaluable data. 'Overall' n=participants with evaluable data; 'Last 3 Months on Study' n=participants with evaluable data and >=6 months on study.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Arm 1: Weekly Prophylaxis
Number analyzed (Participants) | 61
IU/kg
  Overall (n=61) | 46.26 (11.304)
  Last 3 months on study (n=58) | 43.10 (15.395)

9. Secondary Outcome: Average Dosing Interval For the Individualized Interval Prophylaxis Arm
Description: Average dosing interval = sum of days in the included dosing intervals divided by the number of included intervals. Participants could have multiple prophylactic dose interval changes. Prophylactic dosing = from first prophylactic injection received for rFIXFc to the last prophylactic injection on study. Intervals between 2 prophylactic doses separated by a bleed/surgery/PK visit were not included. In Arm 2, the efficacy period (EP) started with date and time of first prophylactic dose following a completed PK sampling period and ended with last dose administered (for prophylaxis or a bleeding episode). The EP was interrupted for all surgical/rehabilitation periods (for both major and minor surgeries).
Time Frame: up to 52 weeks ± 1 week (efficacy period as defined in description)
Population: Full Analysis Set: participants in Arm 2 who received at least 1 dose of rFIXFc with >=6 months on study and evaluable data.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm 2: Individualized Interval Prophylaxis
Number analyzed (Participants) | 26
days
  Overall | 12.53 (2.018) [10.38 to 13.37]
  Last 3 months on study | 14.00 (2.864) [11.29 to 14.00]

10. Secondary Outcome: Annualized Bleeding Rate by Type of Bleed (Spontaneous and Traumatic)
Description: Annualized bleeding episodes = (number of bleeding episodes/number of days in efficacy period)*365.25. Please see the definition of the efficacy period (EP) in the Outcome Measure 4 Description. The EP was interrupted for the repeat PK period in Arm 1 (sequential PK subgroup) and for all surgical/rehabilitation periods (for both major and minor surgeries) in all 3 arms. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered the same bleeding episode. Any bleeding at a different location was a separate bleeding episode regardless of time from the last injection.
Time Frame: up to 52 weeks ± 1 week (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc with evaluable data.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 61 | 26 | 27
episodes per participant per year
  Spontaneous | 1.04 (2.154) [0.00 to 2.19] | 0.88 (1.780) [0.00 to 2.30] | 11.78 (11.096) [2.62 to 19.78]
  Traumatic | 0.99 (1.539) [0.00 to 2.13] | 0.00 (2.065) [0.00 to 0.78] | 2.21 (7.214) [0.00 to 6.81]
  Unknown | 0.00 (0.603) [0.00 to 0.00] | 0.00 (0.705) [0.00 to 0.00] | 0.00 (1.043) [0.00 to 1.34]

11. Secondary Outcome: Annualized Bleeding Rate by Location of Bleed (Joint, Muscle, Internal, Skin/Mucosa)
Description: as for outcome 10
Time Frame: up to 52 weeks ± 1 week (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc with evaluable data.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 61 | 26 | 27
episodes per participant per year
  Joint | 1.11 (2.678) [0.00 to 4.01] | 0.36 (2.498) [0.00 to 3.24] | 13.58 (10.418) [6.13 to 21.61]
  Muscle | 0.00 (1.273) [0.00 to 1.04] | 0.00 (0.902) [0.00 to 0.00] | 3.96 (3.733) [1.02 to 6.79]
  Internal | 0.00 (0.562) [0.00 to 0.00] | 0.00 (0.448) [0.00 to 0.00] | 0.00 (0.893) [0.00 to 1.31]
  Skin/Mucosa | 0.00 (0.668) [0.00 to 0.00] | 0.00 (0.472) [0.00 to 0.00] | 0.00 (2.968) [0.00 to 1.14]

12. Secondary Outcome: Number of Days From Last Injection to Treat a New Bleeding Episode
Description: Please see the definition of the Efficacy Period (EP) in the Outcome Measure 4 Description. The EP was interrupted for the repeat PK period in Arm 1 (sequential PK subgroup) and for all surgical/rehabilitation periods (for both major and minor surgeries) in all 3 arms. A follow-up injection administered >72 hours after the most recent injection given to treat a bleed was considered a new bleed at the same location and was classified as type=Unknown (bleeding episodes of this type were not evaluable). The first bleed for each participant could not be included in this analysis since there was no previous bleed from which to measure time. The number of days from the last injection to treat a bleed to a new bleeding episode was analyzed across all evaluable bleeding episodes per participant.
Time Frame: up to 52 weeks ± 1 week (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc and at least 1 evaluable bleeding episode.
Measure: Median (Inter-Quartile Range); unit: days
Units Other Than Participants: Evaluable Bleeding Episodes
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 35 | 13 | 27
Number analyzed (Evaluable Bleeding Episodes) | 110 | 45 | 359
days
  Per Bleeding Episode | 40.78 (57.184) [14.10 to 78.63] | 39.48 (63.228) [26.05 to 84.82] | 13.42 (21.837) [8.00 to 22.83]
  Per Participant | 59.52 (49.610) [37.39 to 88.78] | 76.13 (37.451) [51.38 to 98.29] | 19.67 (40.576) [15.61 to 32.86]

13. Secondary Outcome: Number of Injections Required for Resolution of a Bleeding Episode
Description: In Arms 1 and 2, the efficacy period (EP) started with date and time of first prophylactic dose following a completed PK sampling period and ended with last dose administered (for prophylaxis or a bleeding episode). In Arm 3, the EP started following last PK sampling timepoint and ended with either date of last contact or date of last entry into the eDiary, whichever was later. The EP was interrupted for the repeat PK period in Arm 1 and for all surgical/rehabilitation periods in all 3 arms. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered the same bleeding episode. All injections given from the initial sign of a bleed until the last date/time within the bleed window are counted. The resolution of a bleed is defined as no sign of bleeding following injection for the bleed.
Time Frame: up to 52 weeks ± 1 week (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc and had at least 1 bleeding episode.
Measure: Median (Inter-Quartile Range); unit: injections
Units Other Than Participants: Bleeding Episodes
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 47 | 15 | 27
Number analyzed (Bleeding Episodes) | 167 | 67 | 402
injections
  Per Bleeding Episode | 1.0 (0.56) [1.0 to 1.0] | 1.0 (0.53) [1.0 to 1.0] | 1.0 (0.31) [1.0 to 1.0]
  Per Participant | 1.00 (0.50) [1.00 to 1.25] | 1.09 (0.30) [1.00 to 1.33] | 1.04 (0.32) [1.00 to 1.08]

14. Secondary Outcome: Number of Injections Required for Resolution of a Bleeding Episode by Location of Bleed
Description: Please see the definition of the efficacy period (EP) in the Outcome Measure 4 Description. The EP was interrupted for the repeat PK period in Arm 1 (sequential PK subgroup) and for all surgical/rehabilitation periods (for both major and minor surgeries) in all 3 arms. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered the same bleeding episode. All injections given from the initial sign of a bleed until the last date/time within the bleed window were counted. The resolution of a bleed was defined as no sign of bleeding following injection for the bleed. Bleeding episodes that presented in multiple locations are included as a single event in the overall summary for the number of injections to resolve that bleeding episode but are included in summaries for each location.
Time Frame: up to 52 weeks ± 1 week (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc, had a bleeding episode, and had evaluable efficacy assessments; n=total number of bleeds at given location.
Measure: Median (Inter-Quartile Range); unit: injections
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 47 | 15 | 27
injections
  Joint (n=125, 52, 314) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Muscle (n=35, 10, 90) | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Internal (n=9, 3, 11) | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Skin/Mucosa (n=11, 4, 21) | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

15. Secondary Outcome: Total Dose Per Injection Required for Resolution of a Bleeding Episode by Location of Bleed
Description: For each bleeding episode at one location, the total dose is the sum of the doses (IU/kg) administered across all injections given to treat that bleeding episode. Please see the definition of the efficacy period (EP) in the Outcome Measure 4 Description. The EP was interrupted for the repeat PK period in Arm 1 (sequential PK subgroup) and for all surgical/rehabilitation periods (for both major and minor surgeries) in all 3 arms. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered the same bleeding episode. Bleeding episodes that presented in multiple locations are included as a single event in the overall summary for dose administered to resolve that bleeding episode but are included in the individual summaries for each location.
Time Frame: up to 52 weeks ± 1 week (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc, had a bleeding episode, and had complete information on the dose administered to treat a bleeding episode; n=total number of bleeding episodes at this location.
Measure: Median (Inter-Quartile Range); unit: IU/kg
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 47 | 15 | 27
IU/kg
  Joint (n=124, 52, 313) | 50.14 [31.65 to 61.64] | 45.29 [35.71 to 97.41] | 46.73 [33.33 to 60.79]
  Muscle (n=35, 10, 90) | 55.56 [46.89 to 88.16] | 67.17 [33.63 to 87.46] | 46.57 [33.33 to 60.79]
  Internal (n=9, 3, 11) | 48.72 [41.67 to 125.00] | 70.26 [33.63 to 131.72] | 46.73 [33.33 to 61.07]
  Skin/Mucosa (n=11, 4, 21) | 46.89 [38.67 to 79.55] | 48.48 [34.50 to 79.69] | 22.22 [20.83 to 36.36]

16. Secondary Outcome: Hemophilia-Specific Quality of Life Index for Adults (Haem-A-QoL) Questionnaire: Change From Baseline to Week 26
Description: The Haem-A-QoL consists of items pertaining to 10 domains specific to living with hemophilia and was administered to adult participants (> 17 years). The areas covered by this instrument are: physical health, feeling, view of yourself, sports/leisure, school/work, dealing with hemophilia, and treatment (all 7 domains, during the last month) and future, family planning, and outlook for the future (all 3 domains, recently). Changes from baseline for the Haem-A-QoL questionnaire are summarized by prestudy treatment regimen (pooled for Arms 1 and 2). Lower scores represent better QoL; therefore, a negative change from baseline represents improvement during the course of the study. Scores on a scale range between 0 and 100.
Time Frame: Baseline, Week 26
Population: Full Analysis Set: participants in the 2 prophylaxis arms (Arms 1 and 2) over 17 years of age who received at least 1 dose of rFIXFc and had an assessment. n=participants who had specified assessment at given timepoint.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Pre-study Regimen: Prophylaxis (Arms 1 and 2 Pooled): Participants from the Weekly or Individualized Interval Prophylaxis Arms (Arms 1 or 2) who had a prophylaxis pre-study regimen.
- Pre-study Regimen: On Demand (Arms 1 and 2 Pooled): Participants from the Weekly or Individualized Interval Prophylaxis Arms (Arms 1 or 2) who had an on-demand pre-study regimen.
Arm/Group | Pre-study Regimen: Prophylaxis (Arms 1 and 2 Pooled) | Pre-study Regimen: On Demand (Arms 1 and 2 Pooled)
Number analyzed (Participants) | 27 | 31
units on a scale
  Total Score (n=27, 26) | -6.82 [-22.8 to 6.1] | -6.25 [-25.5 to 12.8]
  Physical Health (n=27, 31) | -10.00 [-45.0 to 20.0] | -15.00 [-60.0 to 15.0]
  Feeling (n=27, 31) | 0.00 [-43.8 to 50.0] | 0.00 [-43.8 to 62.5]
  View of Yourself (n=27, 30) | -5.00 [-25.0 to 15.0] | -5.00 [-35.0 to 25.0]
  Sports and Leisure (n=22, 21) | -7.50 [-70.0 to 25.0] | -20.0 [-40.0 to 35.0]
  Work and School (n=22, 25) | 0.00 [-31.3 to 52.1] | -6.25 [-31.3 to 18.8]
  Dealing with Hemophilia (n=27, 31) | 0.00 [-100.0 to 100.0] | -8.33 [-66.7 to 75.0]
  Treatment (n=27, 31) | -6.25 [-18.8 to 18.8] | 0.00 [-53.1 to 37.5]
  Future (n=26, 30) | -5.00 [-25.0 to 10.0] | 0.00 [-30.0 to 20.0]
  Family Planning (n=15, 13) | 0.00 [-29.2 to 12.5] | 0.00 [-43.8 to 25.0]
  Partnership and Sexuality (n=26, 30) | 0.00 [-50.0 to 66.7] | 0.00 [-25.0 to 25.0]

17. Secondary Outcome: Haem-A-QoL Questionnaire for Adults: Change From Baseline to Week 52
Description: as for outcome 16
Time Frame: Baseline, Week 52
Population: as for outcome 16
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pre-study Regimen: Prophylaxis (Arms 1 and 2 Pooled) | Pre-study Regimen: On Demand (Arms 1 and 2 Pooled)
Number analyzed (Participants) | 27 | 24
units on a scale
  Total Score (n=25, 19) | -4.35 [-24.4 to 9.6] | -6.06 [-31.0 to 1.0]
  Physical Health (n=26, 23) | -10.00 [-45.0 to 20.0] | -15.00 [-60.0 to 0.0]
  Feeling (n=26, 23) | 0.00 [-37.5 to 75.0] | 0.00 [-50.0 to 18.8]
  View of Yourself (n=26, 24) | -7.50 [-45.0 to 20.0] | -5.00 [-35.0 to 15.0]
  Sports and Leisure (n=20, 16) | -0.62 [-55.0 to 27.5] | -17.50 [-55.0 to 17.5]
  Work and School (n=22, 20) | 0.00 [-31.3 to 25.0] | -3.13 [-41.7 to 25.0]
  Dealing with Hemophilia (n=27, 24) | 0.00 [-66.7 to 33.3] | 4.17 [-66.7 to 66.7]
  Treatment (n=27, 24) | -6.25 [-30.8 to 15.6] | -4.69 [-34.4 to 34.4]
  Future (n=26, 23) | -5.00 [-40.0 to 20.0] | -5.00 [-40.0 to 15.0]
  Family Planning (n=14, 11) | 0.00 [-25.0 to 33.3] | 0.00 [-12.5 to 12.5]

18. Secondary Outcome: Hemophilia-Specific Quality of Life Index for Children (Haemo-QoL) Questionnaire: Change From Baseline to Week 26 and Week 52
Description: The Haemo-QoL, a quality of life (QoL) assessment instrument for children and adolescents with hemophilia, was administered to participants from 13- to 17-years-old. This instrument assesses domains specific to living with hemophilia. For the Haemo-QoL, higher scores indicate a worse quality of life. Scores on a scale range between 0 and 100.
Time Frame: Baseline, Week 26, Week 52
Population: No summary analysis was done for this outcome measure due to the small number of participants completing the questionnaire.
Groups:
- Pre-study Regimen: Prophylaxis (Arms 1 and 2 Pooled): Child and adolescent participants from the Weekly or Individualized Interval Prophylaxis Arms (Arms 1 or 2) who had a prophylaxis pre-study regimen.
- Pre-study Regimen: On Demand (Arms 1 and 2 Pooled): Child and adolescent participants from the Weekly or Individualized Interval Prophylaxis Arms (Arms 1 or 2) who had an on-demand pre-study regimen.
Arm/Group | Pre-study Regimen: Prophylaxis (Arms 1 and 2 Pooled) | Pre-study Regimen: On Demand (Arms 1 and 2 Pooled)
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Investigators'/Surgeons' Assessment of Participants' Response to rFIXFc for Major Surgery
Description: Based on the first assessment of hemostasis by the surgeon/investigator 24 hours or later post-surgery. Scaled responses: Excellent = 1, Good = 2, Fair = 3, Poor/none = 4.
Time Frame: up to 52 weeks ± 1 week
Population: Participants in Arm 4 who received at least 1 dose of rFIXFc.
Measure: Number; unit: responses
Units Other Than Participants: Major Surgeries
Arm/Group | Arm 4: Perioperative Management
Number analyzed (Participants) | 12
Number analyzed (Major Surgeries) | 14
responses
  Excellent or Good | 14
  Excellent | 13
  Good | 1
  Fair | 0
  Poor/None | 0

20. Secondary Outcome: Number of Injections Required to Maintain Hemostasis During Major Surgery
Description: The number of injections to maintain hemostasis during surgery includes all injections for surgery purposes including the loading dose to the end date/time of surgery.
Time Frame: up to 52 weeks ± 1 week
Population: Participants in Arm 4 who received at least 1 dose of rFIXFc.
Measure: Median (Full Range); unit: injections
Units Other Than Participants: Major Surgeries
Arm/Group | Arm 4: Perioperative Management
Number analyzed (Participants) | 12
Number analyzed (Major Surgeries) | 14
injections | 1.00 (0.825) [1.0 to 4.0]

21. Secondary Outcome: Dose Per Injection and Total Dose Required to Maintain Hemostasis During Major Surgery
Description: Mean dose per injection is the average dose for all injections (including loading dose) needed to maintain hemostasis during surgery. Total dose is the sum across all injections (including loading dose) needed to maintain hemostasis during surgery.
Time Frame: up to 52 weeks ± 1 week
Population: Participants in Arm 4 who received at least 1 dose of rFIXFc.
Measure: Median (Full Range); unit: IU/kg
Units Other Than Participants: Major Surgeries
Arm/Group | Arm 4: Perioperative Management
Number analyzed (Participants) | 12
Number analyzed (Major Surgeries) | 14
IU/kg
  Dose per Injection | 90.91 (30.869) [49.4 to 142.3]
  Total Dose | 102.59 (60.930) [49.4 to 264.5]

22. Secondary Outcome: Estimated Total Blood Loss During Major Surgery
Time Frame: up to 52 weeks ± 1 week
Population: Participants in Arm 4 who received at least 1 dose of rFIXFc.
Measure: Median (Full Range); unit: mL
Units Other Than Participants: Major Surgeries
Arm/Group | Arm 4: Perioperative Management
Number analyzed (Participants) | 12
Number analyzed (Major Surgeries) | 14
mL | 65.50 (95.161) [0.0 to 300.0]

23. Primary Outcome: Incidence Rate of FIX Inhibitor Development
Description: An inhibitor test result ≥0.6 Bethesda units (BU)/mL, identified and confirmed by re-testing of a second sample obtained within 2 to 4 weeks, was considered positive. Both tests were to be performed using the Nijmegen-modified Bethesda Assay by the central laboratory. The incidence rates along with the 95% CI were summarized for all titers for subjects with 50 or more exposure days (EDs) to rFIXFc and a valid inhibitor test after the 50th exposure. In addition, the incidence rates for all subjects regardless of their exposure days to rFIXFc were also summarized. The 95% CI was calculated using Clopper-Pearson exact method.
Time Frame: up to 52 weeks ± 1 week
Population: Safety Analysis Set: participants who received at least 1 dose of of rFIXFc and who had a valid inhibitor test; n=number of participants with given number of exposure days who had a valid inhibitor test.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total: All participants from Arms 1-4
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand) | Arm 4: Perioperative Management | Total
Number analyzed (Participants) | 63 | 27 | 27 | 4 | 121
percentage of participants
  Participants with>=50 EDs to rFIXFc(n=52,2,0,1,55) | 0 [0 to 6.85] | 0 [0 to 84.19] | 0 [NA to NA] — n=0 for this arm | 0 [0 to 97.50] | 0 [0 to 6.49]
  All participants (n=63, 27, 27, 4, 121) | 0 [0 to 5.69] | 0 [0 to 12.77] | 0 [0 to 12.77] | 0 [0 to 60.24] | 0 [0 to 3.00]

24. Secondary Outcome: Number of Transfusions Required Per Surgery
Description: Number of blood component transfusions during a single surgery.
Time Frame: up to 52 weeks ± 1 week
Population: Participants in Arm 4 who received at least 1 dose of rFIXFc.
Measure: Number; unit: surgeries
Units Other Than Participants: Major Surgeries
Arm/Group | Arm 4: Perioperative Management
Number analyzed (Participants) | 12
Number analyzed (Major Surgeries) | 14
surgeries
  0 transfusions | 12
  1 transfusion | 0
  2 transfusions | 1
  3 transfusions | 0
  >3 transfusions | 1

25. Secondary Outcome: Maximum Concentration (Cmax)
Description: Maximum concentration during a dosing interval. Assessment of FIX activity with BeneFIX was conducted following a required 120-hour (5-day) washout period, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 72 (±3) hours, and 96 (±3) hours (4 days) from the start of the injection. Assessment of FIX activity and rFIXFc concentration was conducted following the initial dose of rFIXFc (after a required 120-hour [5-day] washout period) and at Week 26, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 96 (±3) hours (4 days), 144 (±3) hours (6 days), 168 (±3) hours (7 days), 192 (±3) hours (8 days), and 240 (±3) hours (10 days) from the start of the injection.
Time Frame: See Measure Description for complete time frame. Each participant was to complete PK sampling up to, and including, the 96-hour (4-day) timepoint for BeneFIX PK assessment and the 240-hour (10-day) timepoint for rFIXFc PK assessment.
Population: Participants in the Sequential PK Subgroup who have evaluable PK profiles for both BeneFIX and baseline rFIXFc.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Groups:
- Arm 1: Weekly Prophylaxis - Sequential PK Subgroup: Prior to the first dose of rFIXFc, participants in the Sequential PK subgroup were to receive a single dose of 50 IU/kg BeneFIX administered IV in the clinic, followed by PK sampling. A single dose of 50 IU/kg rFIXFc was administered following a 120-hour washout from BeneFIX, followed by PK sampling for a baseline PK profiling. At Week 26 (±1 week) subjects were to receive a single dose of 50 IU/kg rFIXFc for repeat PK profiling.
  All participants in Arm 1 received 50 IU/kg rFIXFc via intravenous (IV) injection once every 7 days initially, then at a dose indicated by the participant's baseline pharmacokinetic (PK) assessment that ensured a target trough of 1% to 3% above baseline or higher, as clinically indicated. Adjustments to the initial weekly dose of rFIXFc (50 IU/kg) were to be made based on baseline PK assessments, occurrence of spontaneous bleeding episodes, and the trough levels, which were to be monitored at Weeks 4, 16, 26, and 39.
Arm/Group | Arm 1: Weekly Prophylaxis - Sequential PK Subgroup
Number analyzed (Participants) | 22
IU/dL
  rFIXFc Baseline | 40.81 [33.60 to 49.58]
  BeneFIX | 43.08 [36.69 to 50.59]

26. Secondary Outcome: Area Under the Curve (AUC) Per Dose
Description: Dose normalized area under the drug concentration-time curve. Assessment of FIX activity with BeneFIX was conducted following a required 120-hour (5-day) washout period, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 72 (±3) hours, and 96 (±3) hours (4 days) from the start of the injection. Assessment of FIX activity and rFIXFc concentration was conducted following the initial dose of rFIXFc (after a required 120-hour [5-day] washout period) and at Week 26, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 96 (±3) hours (4 days), 144 (±3) hours (6 days), 168 (±3) hours (7 days), 192 (±3) hours (8 days), and 240 (±3) hours (10 days) from the start of the injection.
Time Frame: as for outcome 25
Population: Participants in the Sequential PK Subgroup who have evaluable PK profiles for both BeneFIX and baseline rFIXFc.
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL per IU/kg
Arm/Group | Arm 1: Weekly Prophylaxis - Sequential PK Subgroup
Number analyzed (Participants) | 22
IU*h/dL per IU/kg
  rFIXFc Baseline | 31.32 [27.88 to 35.18]
  BeneFIX | 15.77 [14.02 to 17.74]

27. Secondary Outcome: Half Life (t1/2) Alpha and t1/2 Beta
Description: Time required for the concentration of the drug to reach half of its original value. Alpha and beta half-life indicate distribution and elimination half-life in a two-compartment PK model. Assessment of FIX activity with BeneFIX was conducted following a required 120-hour (5-day) washout period, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 72 (±3) hours, and 96 (±3) hours (4 days) from the start of the injection. Assessment of FIX activity and rFIXFc concentration was conducted following the initial dose of rFIXFc (after a required 120-hour [5-day] washout period) and at Week 26, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 96 (±3) hours (4 days), 144 (±3) hours (6 days), 168 (±3) hours (7 days), 192 (±3) hours (8 days), and 240 (±3) hours (10 days) from the start of the injection.
Time Frame: as for outcome 25
Population: Participants in the Sequential PK Subgroup who have evaluable PK profiles for both BeneFIX and baseline rFIXFc.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Arm 1: Weekly Prophylaxis - Sequential PK Subgroup
Number analyzed (Participants) | 22
hours
  rFIXFc Baseline: t1/2 alpha | 5.0279 [3.2032 to 7.8919]
  BeneFIX: t1/2 alpha | 2.4113 [1.6183 to 3.5930]
  rFIXFc Baseline: t1/2 beta | 82.12 [71.39 to 94.46]
  BeneFIX: t1/2 beta | 33.77 [29.13 to 39.15]

28. Secondary Outcome: Clearance (CL)
Description: The measure of the efficiency of the body to remove the drug and the unit is the volume of the plasma or blood cleared of drug per unit time. Assessment of FIX activity with BeneFIX was conducted following a required 120-hour (5-day) washout period, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 72 (±3) hours, and 96 (±3) hours (4 days) from the start of the injection. Assessment of FIX activity and rFIXFc concentration was conducted following the initial dose of rFIXFc (after a required 120-hour [5-day] washout period) and at Week 26, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 96 (±3) hours (4 days), 144 (±3) hours (6 days), 168 (±3) hours (7 days), 192 (±3) hours (8 days), and 240 (±3) hours (10 days) from the start of the injection.
Time Frame: as for outcome 25
Population: Participants in the Sequential PK Subgroup who have evaluable PK profiles for both BeneFIX and baseline rFIXFc.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | Arm 1: Weekly Prophylaxis - Sequential PK Subgroup
Number analyzed (Participants) | 22
mL/h/kg
  rFIXFc Baseline | 3.193 [2.843 to 3.587]
  BeneFIX | 6.340 [5.637 to 7.131]

29. Secondary Outcome: Mean Residence Time (MRT)
Description: The average time for all the drug molecules to reside in the body. Assessment of FIX activity with BeneFIX was conducted following a required 120-hour (5-day) washout period, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 72 (±3) hours, and 96 (±3) hours (4 days) from the start of the injection. Assessment of FIX activity and rFIXFc concentration was conducted following the initial dose of rFIXFc (after a required 120-hour [5-day] washout period) and at Week 26, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 96 (±3) hours (4 days), 144 (±3) hours (6 days), 168 (±3) hours (7 days), 192 (±3) hours (8 days), and 240 (±3) hours (10 days) from the start of the injection.
Time Frame: as for outcome 25
Population: Participants in the Sequential PK Subgroup who have evaluable PK profiles for both BeneFIX and baseline rFIXFc.
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Arm 1: Weekly Prophylaxis - Sequential PK Subgroup
Number analyzed (Participants) | 22
hours
  rFIXFc Baseline | 98.60 [88.16 to 110.29]
  BeneFIX | 41.19 [35.98 to 47.15]

30. Secondary Outcome: Volume in Steady State (Vss)
Description: Volume of distribution at steady state. Assessment of FIX activity with BeneFIX was conducted following a required 120-hour (5-day) washout period, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 72 (±3) hours, and 96 (±3) hours (4 days) from the start of the injection. Assessment of FIX activity and rFIXFc concentration was conducted following the initial dose of rFIXFc (after a required 120-hour [5-day] washout period) and at Week 26, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 96 (±3) hours (4 days), 144 (±3) hours (6 days), 168 (±3) hours (7 days), 192 (±3) hours (8 days), and 240 (±3) hours (10 days) from the start of the injection.
Time Frame: as for outcome 25
Population: Participants in the Sequential PK Subgroup who have evaluable PK profiles for both BeneFIX and baseline rFIXFc.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | Arm 1: Weekly Prophylaxis - Sequential PK Subgroup
Number analyzed (Participants) | 22
mL/kg
  rFIXFc Baseline | 314.8 [277.8 to 356.8]
  BeneFIX | 261.1 [222.9 to 305.9]

31. Secondary Outcome: Incremental Recovery
Description: IU/dL rise in plasma per IU/kg drug administered. Assessment of FIX activity with BeneFIX was conducted following a required 120-hour (5-day) washout period, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 72 (±3) hours, and 96 (±3) hours (4 days) from the start of the injection. Assessment of FIX activity and rFIXFc concentration was conducted following the initial dose of rFIXFc (after a required 120-hour [5-day] washout period) and at Week 26, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 96 (±3) hours (4 days), 144 (±3) hours (6 days), 168 (±3) hours (7 days), 192 (±3) hours (8 days), and 240 (±3) hours (10 days) from the start of the injection.
Time Frame: as for outcome 25
Population: Participants in the Sequential PK Subgroup who have evaluable PK profiles for both BeneFIX and baseline rFIXFc.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | Arm 1: Weekly Prophylaxis - Sequential PK Subgroup
Number analyzed (Participants) | 22
IU/dL per IU/kg
  rFIXFc Baseline | 0.9211 [0.7710 to 1.1004]
  BeneFIX | 0.9451 [0.8149 to 1.0961]

32. Secondary Outcome: Time to 1% and 3% FIX Activity
Description: Time to reach 1 or 3 IU/dL (%) after a single dose. Assessment of FIX activity with BeneFIX was conducted following a required 120-hour (5-day) washout period, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 72 (±3) hours, and 96 (±3) hours (4 days) from the start of the injection. Assessment of FIX activity and rFIXFc concentration was conducted following the initial dose of rFIXFc (after a required 120-hour [5-day] washout period) and at Week 26, at these timepoints: predose, 10 (±2) minutes, 1 hour (±15 minutes), 3 hours (±15 minutes), 6 hours (±15 minutes), 24 (±2) hours, 48 (±2) hours, 96 (±3) hours (4 days), 144 (±3) hours (6 days), 168 (±3) hours (7 days), 192 (±3) hours (8 days), and 240 (±3) hours (10 days) from the start of the injection.
Time Frame: as for outcome 25
Population: Participants in the Sequential PK Subgroup who have evaluable PK profiles for both BeneFIX and baseline rFIXFc.
Measure: Geometric Mean (95% Confidence Interval); unit: days
Arm/Group | Arm 1: Weekly Prophylaxis - Sequential PK Subgroup
Number analyzed (Participants) | 22
days
  rFIXFc Baseline: 1% Activity | 11.224 [10.200 to 12.350]
  BeneFIX: 1% Activity | 5.087 [4.579 to 5.651]
  rFIXFc Baseline: 3% Activity | 5.767 [5.066 to 6.565]
  BeneFIX: 3% Activity | 2.832 [2.568 to 3.123]

33. Secondary Outcome: Number of Participants With Clinically Relevant Abnormalities or Relevant Changes From Baseline in Vital Signs
Description: Number of participants with clinically relevant abnormalities or relevant changes from baseline in temperature, pulse (beats per minute [bpm]), systolic blood pressure (SBP), and diastolic blood pressure (DBP) are presented. Baseline (BL) is defined as the last non-missing evaluable assessment taken prior and closest to the first rFIXFc dose. Because the perioperative management period represents a unique clinical situation, safety data obtained during the surgical/rehabilitation period for participants in Arm 4 were included in listings and reviewed separately. Review of the listing was sufficient to assess this endpoint.
Time Frame: up to 52 weeks ± 1 week
Population: Safety Analysis Set: participants who received at least 1 dose of BeneFIX or rFIXFc; a table was not generated for participants in the perioperative management/surgical arm (Arm 4). n=participants with a baseline assessment and at least one post-baseline assessment for temperature or at least one post-baseline assessment for pulse, SBP, and DBP.
Measure: Number; unit: participants
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 63 | 29 | 27
participants
  Temperature: >38°C and ≥1°C ↑ from BL, n=61,28,24 | 0 | 0 | 0
  Pulse: >120 bpm or >20 bpm ↑ from BL, n=62,28,24 | 1 | 2 | 0
  Pulse: <50 bpm or >20 bpm ↓ from BL, n=62,28,24 | 2 | 1 | 0
  SBP: >180 mm Hg or >40 mm Hg ↑ from BL, n=62,28,24 | 0 | 1 | 0
  SBP: <90 mm Hg or >30 mm Hg ↓ from BL, n=62,28,24 | 4 | 1 | 0
  DBP: >105 mm Hg or >30 mm Hg ↑ from BL, n=62,28,24 | 3 | 0 | 0
  DBP: <50 mm Hg or >20 mm Hg ↓ from BL, n=62,28,24 | 5 | 4 | 0

34. Secondary Outcome: Coagulation Parameter: Change From Pre-dose Values in Prothrombin Split Fragments 1+ 2 (F 1+2)
Description: Maximum value post-dosing is defined as maximum value over the 1-, 6-, and 24-hour evaluations.
Time Frame: Pre-dose, 1 hour post-dose, 6 hours post-dose, and 24 hours post-dose at baseline (120 hours before Day 1, for BeneFIX), Day 1, Week 26, and Week 52 (for rFIXFc)
Population: The Sequential PK subgroup consisted of all participants who had evaluable PK profiles for both BeneFIX and baseline rFIXFc, and/or evaluable PK profiles for both baseline and repeat rFIXFc at Week 26 (±1 week). n=participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- Sequential PK Subgroup: BeneFIX; Sequential PK Subgroup: rFIXFc Day 1; Sequential PK Subgroup: rFIXFc Week 26; Sequential PK Subgroup: rFIXFc Week 52: Prior to the first dose of rFIXFc, participants in the Sequential PK subgroup were to receive a single dose of 50 IU/kg BeneFIX administered IV in the clinic, followed by PK sampling. A single dose of 50 IU/kg rFIXFc was administered following a 120-hour washout from BeneFIX, followed by PK sampling for a baseline PK profiling. At Week 26 (±1 week) subjects were to receive a single dose of 50 IU/kg rFIXFc for repeat PK profiling.
  All participants in Arm 1 received 50 IU/kg rFIXFc via intravenous (IV) injection once every 7 days initially, then at a dose indicated by the participant's baseline PK assessment that ensured a target trough of 1% to 3% above baseline or higher, as clinically indicated. Adjustments to the initial weekly dose of rFIXFc (50 IU/kg) were to be made based on baseline PK assessments, occurrence of spontaneous bleeding episodes, and the trough levels, which were to be monitored at Weeks 4, 16, 26, and 39.
Arm/Group | Sequential PK Subgroup: BeneFIX | Sequential PK Subgroup: rFIXFc Day 1 | Sequential PK Subgroup: rFIXFc Week 26 | Sequential PK Subgroup: rFIXFc Week 52
Number analyzed (Participants) | 23 | 23 | 23 | 23
pmol/L
  Pre-dosing Value (n=23, 23, 20, 19) | 134.1 (64.93) | 130.0 (57.55) | 131.6 (42.43) | 176.7 (112.36)
  Change at 1 Hour Post-dosing (n=23, 22, 20, 0) | 73.4 (171.68) | 8.6 (39.14) | 1.3 (51.64) | NA (NA) — assessment was not done at this time point
  Change at 6 Hours Post-dosing (n=23, 22, 20, 0) | 7.8 (55.45) | 8.3 (38.66) | -4.4 (45.95) | NA (NA) — assessment was not done at this time point
  Change at 24 Hours Post-dosing (n=23, 22, 18, 0) | -3.7 (34.39) | 9.8 (45.62) | 1.7 (27.14) | NA (NA) — assessment was not done at this time point
  Maximum Post-dosing Change (n=23, 23, 19, 0) | 83.0 (168.71) | 30.9 (48.52) | 20.4 (49.38) | NA (NA) — assessment was not done at this time point

35. Secondary Outcome: Coagulation Parameter: Change From Pre-dose Values in Thrombin-antithrombin (TAT) Complex
Description: Maximum value post-dosing is defined as maximum value over the 1-, 6-, and 24-hour evaluations.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sequential PK Subgroup: BeneFIX | Sequential PK Subgroup: rFIXFc Day 1 | Sequential PK Subgroup: rFIXFc Week 26 | Sequential PK Subgroup: rFIXFc Week 52
Number analyzed (Participants) | 23 | 23 | 23 | 23
ng/mL
  Pre-dosing Value (n=23, 23, 20, 19) | 2.87 (2.891) | 2.87 (2.230) | 3.11 (4.075) | 4.28 (7.588)
  Change at 1 Hour Post-dosing (n=23, 22, 20, 0) | 6.67 (15.491) | 1.05 (4.019) | 0.11 (5.813) | NA (NA) — assessment was not done at this time point
  Change at 6 Hours Post-dosing (n=23, 22, 20, 0) | 1.91 (7.303) | 1.07 (4.686) | -0.09 (5.763) | NA (NA) — assessment was not done at this time point
  Change at 24 Hours Post-dosing (n=23, 22, 18, 0) | -0.58 (2.968) | 0.81 (6.095) | -1.10 (4.308) | NA (NA) — assessment was not done at this time point
  Maximum Post-dosing Change (n=23, 23, 19, 0) | 7.42 (15.416) | 3.63 (7.000) | 0.32 (5.969) | NA (NA) — assessment was not done at this time point

36. Secondary Outcome: Coagulation Parameter: Change From Pre-dose Values in D-dimer
Description: Maximum value post-dosing is defined as maximum value over the 1-, 6-, and 24-hour evaluations.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sequential PK Subgroup: BeneFIX | Sequential PK Subgroup: rFIXFc Day 1 | Sequential PK Subgroup: rFIXFc Week 26 | Sequential PK Subgroup: rFIXFc Week 52
Number analyzed (Participants) | 23 | 23 | 23 | 23
ng/mL
  Pre-dosing Value (n=23, 22, 20, 19) | 153.0 (119.37) | 176.2 (165.48) | 120.5 (73.38) | 134.7 (151.36)
  Change at 1 Hour Post-dosing (n=23, 21, 20, 0) | 35.9 (101.80) | 89.6 (509.24) | -5.9 (28.18) | NA (NA) — assessment was not done at this time point
  Change at 6 Hours Post-dosing (n=23, 21, 20, 0) | 47.6 (259.70) | -39.6 (134.42) | -9.4 (16.84) | NA (NA) — assessment was not done at this time point
  Change at 24 Hours Post-dosing (n=23, 21, 18, 0) | 20.0 (85.93) | -31.0 (138.22) | -8.2 (26.06) | NA (NA) — assessment was not done at this time point
  Maximum Post-dosing Change (n=23, 22, 19, 0) | 95.7 (266.98) | 100.6 (494.70) | 4.8 (16.10) | NA (NA) — assessment was not done at this time point

37. Primary Outcome: Annualized Bleeding Rate
Description: Annualized bleeding episodes = (number of bleeding episodes / number of days in the respective period)*365.25. In Arms 1 and 2, the efficacy period (EP) started with date and time of first prophylactic dose following a completed pharmacokinetic (PK) sampling period and ended with last dose administered (for prophylaxis or a bleeding episode). In Arm 3, the EP started following last PK sampling timepoint and ended with either date of last contact or date of last entry into the eDiary, whichever was later. The EP was interrupted for the repeat PK period in Arm 1 (sequential PK subgroup) and for all surgical/rehabilitation periods (for both major and minor surgeries) in all 3 arms. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered the same bleeding episode.
Time Frame: up to 52 weeks ± 1 week (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 61 | 26 | 27
episodes per participant per year | 2.95 [1.01 to 4.35] | 1.38 [0.00 to 3.43] | 17.69 [10.77 to 23.24]

38. Primary Outcome: Comparison of Annualized Bleeding Rates
Description: Estimated with a factor for arm, based on whole study duration for all participants. Annualized bleeding episodes = (number of bleeding episodes / number of days in the respective period)*365.25. In Arms 1 and 2, the efficacy period (EP) started with date and time of first prophylactic dose following a completed PK sampling period and ended with last dose administered (for prophylaxis or a bleeding episode). In Arm 3, the EP started following last PK sampling timepoint and ended with either date of last contact or date of last entry into the eDiary, whichever was later. The EP was interrupted for the repeat PK period in Arm 1 and for all surgical/rehabilitation periods in all 3 arms. A bleeding episode started from the first sign of a bleed, and ended 72 hours after the last treatment for the bleeding, within which any symptoms of bleeding at the same location, or injections less than or equal to 72 hours apart, were considered the same bleeding episode.
Time Frame: up to 52 weeks ± 1 week (efficacy period as defined in description)
Population: Full Analysis Set: participants who received at least 1 dose of rFIXFc.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Number analyzed (Participants) | 61 | 26 | 27
episodes per participant per year | 3.12 [2.46 to 3.95] | 2.40 [1.67 to 3.47] | 18.67 [14.01 to 24.89]
Statistical Analysis 1: Comparison: Arm 1: Weekly Prophylaxis vs Arm 3: Episodic (On Demand); The null hypothesis for the primary endpoint is no difference between any prevention regimen and the on-demand regimen. The sample size of this study was mainly based on clinical rather than statistical considerations. However it was projected to have > 95% power at the 2-sided 0.05 level of significance, based upon this hypothesis test; Test type: Superiority or Other; p < 0.001, negative binomial model — A hierarchical approach was applied to the comparison of the annualized bleeding rates between the prophylaxis arms and the episodic arm; Bleeding Rate Ratio = 0.17, 95% CI 2-sided [0.11 to 0.24]
Statistical Analysis 2: Comparison: Arm 2: Individualized Interval Prophylaxis vs Arm 3: Episodic (On Demand); The null hypothesis for the primary endpoint is no difference between any prevention regimen and the on-demand regimen. The sample size of this study was mainly based on clinical rather than statistical considerations; Test type: Superiority or Other; p < 0.001, negative binomial model — [p-value comment as in outcome 38, analysis 1]; Bleeding Rate Ratio = 0.13, 95% CI 2-sided [0.08 to 0.20]

ADVERSE EVENTS:
Time Frame: up to 52 weeks + 30 days ± 1 week
Description: As the perioperative management period represents a unique clinical situation, safety data obtained during the surgical/rehabilitation period for Arm 4 subjects were analyzed separately per the Analysis Plan, and not included within the Arms 1-3 analysis. See Outcome Measures 3 and 4 for AE/SAE data for the surgical/rehabilitation period, Arm 4.
Arm/Group | Arm 1: Weekly Prophylaxis | Arm 2: Individualized Interval Prophylaxis | Arm 3: Episodic (On Demand)
Serious Adverse Events (participants affected / at risk) | 5/63 | 4/29 | 4/27
Other Adverse Events (participants affected / at risk) | 29/63 | 17/29 | 11/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Weekly Prophylaxis (N=63) | Arm 2: Individualized Interval Prophylaxis (N=29) | Arm 3: Episodic (On Demand) (N=27)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Weekly Prophylaxis (N=63) | Arm 2: Individualized Interval Prophylaxis (N=29) | Arm 3: Episodic (On Demand) (N=27)
Nasopharyngitis (Infections and infestations) | 13 | 4 | 1
Influenza (Infections and infestations) | 5 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 1
Sinusitis (Infections and infestations) | 3 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 2 | 0
Headache (Nervous system disorders) | 2 | 2 | 2
Dizziness (Nervous system disorders) | 3 | 2 | 0
Weight increased (Investigations) | 1 | 0 | 2
Hypertension (Vascular disorders) | 3 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Allergy to arthropod bite (Immune system disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.